CLINICAL TRIAL: NCT06667440
Title: Effectiveness of Cryotherapy in Nulliparous Women with Dysmenorrhea. a Randomized Controlled Trial
Brief Title: Cryotherapy in Nulliparous Women with Dysmenorrhea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, ESTHER DIAZ-MOHEDO, Profesor Titular, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEUMA: 87-2024-H
Record Dates: First submitted 2024-09-10; First posted 2024-10-31 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-09

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRIOTHERAPY (Experimental): Women in the intervention group will apply cryotherapy on their hypogastrium with a coldpack
  Interventions: Other: Cryotherapy
- CONTROL (No Intervention)

INTERVENTIONS:
Other: Cryotherapy — Women in the intervention group will apply cryotherapy on their hypogastrium with a coldpack
  Arms: CRIOTHERAPY

SUMMARY:
The aim of this randomized controlled trial is to observe the effectiveness of cryotherapy application in nulliparous women with primary dysmenorrhea regarding pain intensity, sleep quality and quality of life. It is also intended to analyse whether the levels of physical activity and the socioeconomic status of the participants are determining factors.

DETAILED DESCRIPTION:
For the recruitment of participants (whose minimum n will be calculated using the G*Power computer software) an online dissemination campaign will be carried out through social networks, physiotherapists specialised in pelvic floor dysfunctions and gynaecologists will be contacted to inquire about the availability of patients who can participate, and students from both the University of Malaga and the University of Valencia will be contacted through official communication channels.

Nulliparous women with primary dysmenorrhea who meet the following inclusion criteria will be recruited: (1) Menstrually active women between the ages of 18 (to avoid guardian authorizations) and 45 (age of onset of menopause according to the National Institute of Aging ), (2) Menstrual cycles ranging from 24 to 38 days according to OASH , (3) Menstrual periods of 3 to 7 days, and (4) Pain lasting 1 to 3 days. Women with a history of underlying diseases causing secondary dysmenorrhea, women with systemic and/or psychiatric illnesses, and women with a history of use of hormonal medications, oral contraceptive pills, or intrauterine devices will be excluded.

The intervention will consist of applying a cold pack to the hypogastric region, with the participant lying supine, twice daily for the first three days of menstruation. Participants will be required to keep an application calendar where they will note when they have applied the cold pack, and will record the variables of interest for this study before and after its application. Three menstrual cycles will be monitored, where researchers responsible for the research team will periodically contact the participants to ensure adherence to the treatment. Participants randomized to the control group will not undergo intervention during this period.

For the dependent variables; pain intensity assessed by the Visual Analogue Scale, sleep quality assessed by the Pittsburgh Sleep Quality Index and quality of life assessed by the World Health Organization Quality of Life Brief Version questionnaire, a statistical analysis will be performed using the repeated measures ANOVA test to determine the evolution of these variables during the three menstrual cycles. A posteriori, a correlation analysis will be performed between the results of this test and the physical activity levels of the participants, assessed using the International Physical Activity Questionnaire-Short Form , in addition to the socioeconomic status, assessed using the Kuppuswamy Socioeconomic Status Scale .

ELIGIBILITY:
Inclusion Criteria:

* Menstrually active women
* Menstrual cycles that vary between 24 and 38 days according to the OASH
* menstrual periods between 3 and 7 days, and
* Pain lasting from 1 to 3 days

Exclusion Criteria:

* Patients suffering diseases that generate secondary dysmenorrhea, with systemic or psychiatric diseases, and patients with a history of use of hormonal medication, birth control pill, or intrauterine devices

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
NUMERICAL RATING SCALE (NRS) | From enrollment to the end of the treatment at 6 months
  Subjective measure used to assess the intensity of pain or other symptoms on a scale from 0 to 10, where 0 indicates no pain or symptom and 10 represents the worst possible experience.
  Interpretation: Higher scores indicate greater severity, allowing clinicians to evaluate changes in symptoms over time or the effectiveness of interventions.

SECONDARY OUTCOMES:
Pittsburgh Quality Sleep Index (PQSI) | From enrollment to the end of the treatment at 6 months
  Self-report questionnaire that assesses sleep quality and disturbances over the past month. It comprises several components, including sleep duration, sleep disturbances, and overall sleep quality.
  Interpretation: Score Range (0-21): 0 indicates no difficulty and higher total score (21) indicates poorer sleep quality, making it useful for identifying individuals with sleep issues and monitoring changes following interventions.
World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | From enrollment to the end of the treatment at 6 months
  Quality of life assessment tool that evaluates an individual's perception of their position in life across four domains: physical health, psychological health, social relationships, and environment.
  Interpretation: Score Range (4-20): Higher scores in each domain reflect better quality of life, helping to identify areas needing improvement and assess the impact of health interventions.

OTHER OUTCOMES:
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | Prior to initiation of treatment
  Questionnaire that measures the level of physical activity in adults over the past week, capturing activities across different intensities (vigorous, moderate, walking).
  Interpretation: Expressed as MET-min per week: . The results help classify individuals as physically active (at least 3000 MET-minutes/week), minimally active (at least 600 MET-min/week), or inactive, informing public health strategies and individual health planning.
Kuppuswamy Socioeconomic Status Scale | Prior to initiation of treatment
  This scale assesses socioeconomic status based on education, occupation, and income. It categorizes individuals into different socioeconomic classes (upper, middle, lower) based on these criteria.
  Interpretation: Score Range (1-29): According to the total score thus calculated, the family is placed in the appropriate socioeconomic class (from 26-29: Upper class to below 5: lower). It provides insights into the social determinants of health and can help correlate socioeconomic factors with health outcomes, aiding in targeted interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaga, Málaga, MALAGA, Spain

IPD SHARING:
Plan to Share IPD: No